CLINICAL TRIAL: NCT04445571
Title: Surfactant Administration by Insure or Thin Catheter
Acronym: SAINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kajsa Bohlin, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180367
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: RDS of Prematurity; Surfactant Deficiency Syndrome Neonatal; Analgesia
Keywords: LISA (Less invasive surfactant administration); INSURE; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Pulmonary Atelectasis; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INSURE (Active Comparator): Surfactant administration by Intubation-surfactant-extubation to CPAP according to standard protocol including premedication with analgesia and sedation.
  Interventions: Procedure: Thin catheter technique or standard ET-tube for surfactant administration
- LISA (Active Comparator): Surfactant administration by thin catheter during spontaneous breathing and continued CPAP according to set protocol including premedication with analgesia.
  Interventions: Procedure: Thin catheter technique or standard ET-tube for surfactant administration

INTERVENTIONS:
Procedure: Thin catheter technique or standard ET-tube for surfactant administration — Surfactant administration by intubation with regular ET-tube followed by immediate extubation to CPAP (INSURE) or by thin catheter during spontaneous breathing and continued CPAP.

SUMMARY:
This trial evaluates the efficacy and safety of surfactant administration with thin catheter technique together with analgesic premedication in comparison with the established INSURE-strategy. It will provide valuable knowledge to improve clinical methodology and enhance lung protective treatment strategies for preterm infants.

DETAILED DESCRIPTION:
To compare two approaches for surfactant administration during CPAP in preterm infants, the INSURE and the LISA technique, using premedication intubation protocols, and investigate aspects of safety, stress and pain, timely administration of the drug, response in oxygenation and pulmonary outcome.

Our study asks whether (P) among infants born <32 weeks' gestation with RDS (I) does surfactant administration with LISA and analgesia premedication (C) versus surfactant administration according to the INSURE protocol (O) improve oxygenation and reduce the rate of respiratory failure and need for intubation and mechanical ventilation (T) within 48 hours of the procedure

Primary outcomes:

1. Positive effect: Oxygenation measured as arterial to alveolar ratio (a/A ratio) at 24 hours post-procedure.
2. Negative effect: Need for mechanical ventilation (MV) within 48 hours post-procedure.

Safety outcomes:

1. Time from meeting the FiO2 or a/A ratio criteria for surfactant treatment until surfactant administration
2. Number of tries before successful intubation/placement of catheter
3. Positive pressure ventilation during the procedure - yes/no/duration (minutes)
4. Stress and pain (changes in heart rate, blood pressure and BIIP-scale)

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 32 completed weeks of gestation on CPAP, with clinical and radiological signs of RDS and need for surfactant treatment.

Exclusion Criteria:

* Infants requiring surfactant as part of delivery room resuscitation are not eligible.

Infants will be excluded from the final analysis if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation, including: congenital diaphragmatic hernia; tracheo-oesophageal fistula or cyanotic heart disease.

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | 24 hours post-procedure
  Arterial to alveolar ratio (a/A ratio)
Mechanical ventilation | 48 hours post-procedure
  Need for intubation and mechanical ventilation (MV)

SECONDARY OUTCOMES:
Duration of ventilatory support | Discharge
  Duration of MV (hours), CPAP (days), Oxygen (days)
Complications | Discharge
  Incidence of air leaks, bronchopulmonary dysplasia, Systemic hypotension, retinopathy, necrotizing entercolitis, intraventricular hemorrhage, persistent duct
Mortality | Discharge
  Death or composite outcome death/BPD
Length of stay | Discharge
  Number of days in NICU and total in neonatal care, including home care

OTHER OUTCOMES:
Delay time | 24 hours
  Time from meeting the FiO2 or a/A ratio criteria for surfactant treatment until surfactant administration
Intubation attempts | 24 hours
  Number of tries before successful intubation/placement of catheter
PPV | 24 hours
  Positive pressure ventilation during the procedure - yes/no/duration (minutes)
Stress and pain | 24 hours
  Changes in heart rate, blood pressure and BIIP-scales

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No